CLINICAL TRIAL: NCT05760040
Title: The Effect of Virtual Reality Application on Pain, Anxiety and Satisfaction of Patients During Intrauterine Device (Iud) Insertion
Brief Title: The Effect of Virtual Reality Application on Pain, Anxiety and Satisfaction of Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Nurdan Demirci, PhD RN, Professor, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MarmaraU-OZ-2023
Record Dates: First submitted 2023-02-25; First posted 2023-03-08 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Pain; Anxiety; Satisfaction
Keywords: Intrauterine device; Virtual Reality; pain; anxiety; satisfaction
MeSH Terms: conditions — Pain; Anxiety Disorders; Personal Satisfaction | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (VR) (Experimental): During the intrauterine device application, 40 women who were included in the virtual reality group will be put on virtual reality glasses and watched the video.
  Interventions: Other: vırtual reality
- Control group (Experimental): Routine hospital protocol will be applied to 40 women included in the control group while intrauterine device application is being made.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: vırtual reality — During the intrauterine device application, 40 women who were included in the virtual reality group will be put on virtual reality glasses and watched the video.
  Arms: Virtual Reality (VR)
Other: Control Group — Routine hospital protocol will be applied to 40 women included in the control group while intrauterine device application is being made.
  Arms: Control group

SUMMARY:
Today, common and easily accessible android-based smart devices capable of running virtual reality are used. The image is obtained using a combination of framed simple optical lenses that hold the phone at a fixed distance perpendicular to the user's gaze direction. The working system of three-dimensional resuscitation devices is based on stereographic vision properties. After the relevant applications are installed on the smartphone, the device divides the screen into two, and thanks to the acquisition of different images for the right and left eyes, the illusion of the spatial existence of three-dimensional animated objects is obtained.

The use of virtual reality application, which is used as a non-pharmacological method in different studies, has not been found in IUD (Intrauterine device) applications. This study was planned to examine the effect of virtual reality applications, which will distract their attention during the procedure, on the pain and anxiety levels experienced in women who underwent IUD in the septic area in Esenyurt Necmi Kadıoğlu State Hospital.

DETAILED DESCRIPTION:
Virtual Reality, which is a type of computer system using human-machine interfaces, has been used in pain and anxiety management in different applications in many areas known as painful medical procedures in recent years. According to the researchers' hypotheses, Virtual Reality acts as a non-pharmacological method, using cognitive and attentional processes on the body's complex pain modulation system. Although the neurobiological mechanisms have not been fully explained in studies, it has been reported that virtual reality applications have positive results in pain management. When patients feel that they are in the image, their attention is effectively distracted from the pain. Thus, the existing perception of pain decreases.

In recent years, virtual reality as a distraction application has been used in clinical medical care to relieve pain. Virtual Reality applications; There are studies showing its effectiveness in pain and anxiety management in many areas such as burn debridement, injection applications, wound care, toothache, endoscopy procedure, phantom and chronic pain, and chemotherapy applications.

The use of virtual reality application, which is used as a non-pharmacological method in different studies, has not been found in IUD (Intrauterine device) applications. This study was planned to examine the effect of virtual reality applications, which will distract their attention during the procedure, on the pain and anxiety levels experienced in women who underwent IUD in the septic area in Esenyurt Necmi Kadıoğlu State Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Not having any psychiatric disease,
* Having no vision, hearing and perception problems,
* At least primary school graduate,
* Can read and write Turkish,
* Hemodynamically stable,
* No previous experience of intrauterine device application women

Exclusion Criteria:

* Under 18 years old,
* Having any psychiatric disease,
* Having vision, hearing and perception problems,
* Illiterate,
* Hemodynamically unstable,
* Women who have had an intrauterine device before

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — women who underwent intrauterine device application
Enrollment: 80 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Visual Analoque Scale =VAS | The VAS is a 100 mm (10 cm) ruler that can be used horizontally or vertically. The value "0" at the beginning level defines painlessness, and the value "10" at the end level defines the most severe pain
  pain

SECONDARY OUTCOMES:
State-Trait-Anxiety-Inventory | The inventory is designed using a 4-point Likert scale. There are ten items in the State-Trait Anxiety Scale.
  Anxiety

OTHER OUTCOMES:
Patient Satisfaction Scale | It is a form consisting of Likert-type questions to determine the satisfaction levels of women prepared by the researchers in line with the literature.
  satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: tuğba öz, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
can be shared after the publication of the article.

REFERENCES:
- [Background] Ford CG, Manegold EM, Randall CL, Aballay AM, Duncan CL. Assessing the feasibility of implementing low-cost virtual reality therapy during routine burn care. Burns. 2018 Jun;44(4):886-895. doi: 10.1016/j.burns.2017.11.020. Epub 2018 Jan 2. PMID 29305105
- [Background] Frey DP, Bauer ME, Bell CL, Low LK, Hassett AL, Cassidy RB, Boyer KD, Sharar SR. Virtual Reality Analgesia in Labor: The VRAIL Pilot Study-A Preliminary Randomized Controlled Trial Suggesting Benefit of Immersive Virtual Reality Analgesia in Unmedicated Laboring Women. Anesth Analg. 2019 Jun;128(6):e93-e96. doi: 10.1213/ANE.0000000000003649. PMID 31094789
- [Background] Guo C, Deng H, Yang J. Effect of virtual reality distraction on pain among patients with hand injury undergoing dressing change. J Clin Nurs. 2015 Jan;24(1-2):115-20. doi: 10.1111/jocn.12626. Epub 2014 Jun 4. PMID 24899241
- [Background] Jin W, Choo A, Gromala D, Shaw C, Squire P. A Virtual Reality Game for Chronic Pain Management: A Randomized, Controlled Clinical Study. Stud Health Technol Inform. 2016;220:154-60. PMID 27046570
- [Background] Pourmand A, Davis S, Marchak A, Whiteside T, Sikka N. Virtual Reality as a Clinical Tool for Pain Management. Curr Pain Headache Rep. 2018 Jun 15;22(8):53. doi: 10.1007/s11916-018-0708-2. PMID 29904806
- [Background] Matheve T, Bogaerts K, Timmermans A. Virtual reality distraction induces hypoalgesia in patients with chronic low back pain: a randomized controlled trial. J Neuroeng Rehabil. 2020 Apr 22;17(1):55. doi: 10.1186/s12984-020-00688-0. PMID 32321516
- [Background] Won AS, Tataru CA, Cojocaru CM, Krane EJ, Bailenson JN, Niswonger S, Golianu B. Two Virtual Reality Pilot Studies for the Treatment of Pediatric CRPS. Pain Med. 2015 Aug;16(8):1644-7. doi: 10.1111/pme.12755. Epub 2015 Apr 30. No abstract available. PMID 25930099